CLINICAL TRIAL: NCT06144229
Title: Real-world Effectiveness of HPV Vaccine in Women Living With HIV and Its Impact on Cervical Cancer Screening Accuracies (LiVes LLC Study)
Brief Title: Real-world Effectiveness of HPV Vaccine in Women Living With HIV and Its Impact on Cervical Cancer Screening Accuracies
Acronym: LiVes-LLC
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Frontier Science & Technology Research Foundation, Inc. (Industry); Albert Einstein College of Medicine (Other); Boston Children's Hospital (Other); St. Jude Children's Research Hospital (Other); University of Colorado, Denver (Other); Bronx-Lebanon Hospital Center Health Care System (Other); University of Miami (Other); Baylor College of Medicine (Other); Children's Hospital New Orleans, LA (Other); Jacobi Medical Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Anna-Barbara Moscicki, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: PH700
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-11

CONDITIONS: Hiv; Hpv
Keywords: HPV vaccine effectiveness among those living with HIV; Biomarker evaluation for triage of primary HPV cervical cancer screening.
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical vaginal normal saline washes Exfoliated cervical cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Self-Collection HPV testing kit from Abbott — Self-swab collection kits, participates will self-collected vaginal swab for hrHPV test (at home or in the clinic)

SUMMARY:
This study will examine both Human papillomavirus (HPV) vaccine effectiveness and Primary high-risk HPV PHS screening triage strategies in women living with HIV (WLHIV) by partnering with the Pediatric HIV/AIDs Cohort Study (PHACS) led, in part, by our investigative team. Among WWH, the study will examine the effectiveness of the HPV vaccine The study will screen approximately 810 WWH using a self-sampling kit and those who are PHS[+] will attend a clinical visit to have colposcopy/biopsy and 4 triage tests. WWH with <CIN 2+ are asked to return annually for colposcopy and HPV genotyping for up to 3 yrs. WWH PHS[-] will be asked to return in Year 2 for rescreening. Those PHS[+] will be followed as above and PHS[-] will be asked to obtain self-collected vaginal samples for HPV genotyping annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age and less than or equal to 40 years of age;
* WLHIV regardless of mode of transmission or HPV vaccination status;
* Current enrollment in the Pediatric HIV/AIDS Cohort Study (PHACS),Surveillance Monitoring for ART Toxicities (SMARTT), Adolescent Master Protocol for Participants 18 Years of Age and Older (AMP Up), Adolescent Master Protocol for Participants 18 Years of Age and Older - Lite (AMP Up Lite), or Health Outcomes around Pregnancy and Exposure to HIV/ARVs (HOPE) studies;
* Willing to participate and able to provide informed consent;
* Willing to grant access to other PHACS/HOPE data; and
* Willing to provide access to medical records.

Exclusion Criteria:

* Currently known to be pregnant via self-report at hrHPV screening for initial consent;
* Special consideration: Women who test positive on urine pregnancy test at the baseline colposcopy visit will be asked to defer their colposcopy until after 6 weeks following the end of the pregnancy. However, pregnancy during follow-up will be allowed, and guidelines for endocervical curettage (ECC) and treatment will be followed.39
* Women known to have active CIN 2 or greater, undergoing active surveillance with colposcopy (per participant report);
* Women with known bleeding disorders;
* Women unable to consent for themselves; and
* Women with a hysterectomy with removal of the cervix will be excluded from the study and, if such a procedure is conducted during the participant's study enrollment, the individual will be censored from analysis at the last visit prior to the hysterectomy and taken off-study.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Approximately 810 WLHIV greater than or equal to 21 years of age to less than or equal to 40 years of age who are current participants in PHACS (SMARTT, AMP Up, and AMP Up Lite) or HOPE will be tested for hrHPV using a Food and Drug Administration (FDA)-approved primary hrHPV screening test from self-collected specimens.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of HPV vaccine in WLHIV | 3-year
  -3-year cumulative risk of (i) vaccine-hrHPV types that persist 12 months or longer, and (ii) histologic (h) CIN 2+ (CIN 2+ throughout the protocol means "CIN 2 and worse").

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Barbara Moscicki, MD, Principal Investigator — University of California, Los Angeles; Denise L Jacobson, PhD,MPH, Study Chair — Harvard School of Public Health (HSPH); Howard D Strickler, MD, MPH, Study Chair — Albert Einstein College of Medicine; Tzy-Jyun Yao, PhD, Study Chair — Harvard School of Public Health (HSPH)
Locations (9):
- United States (9):
  - University of Colorado, Denver, Colorado
  - Univeristy of Miami, Miami, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Bronx-Lebanon Hospital Center Health Care System, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - St. Jude Children's research hospital, Memphis, Tennessee
  - Baylor college of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No